CLINICAL TRIAL: NCT02825836
Title: Phase I/II, First in Human, Dose Escalation Trial of TL 895 Monotherapy in Subjects With Relapsed/Refractory B Cell Malignancies and Expansion of TL-895 Monotherapy and Combination Therapy With Navtemadlin in Treatment-Naïve Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Subjects and Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia or Relapsed/Refractory Small Lymphocytic Lymphoma
Brief Title: Phase I/II, FIH, Dose Escalation Trial of TL-895 and Expansion of TL-895 Monotherapy and Combination Therapy With Navtemadlin in Tx-Naïve and R/R CLL/SLL Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS200662_0001; 2016-000286-23 (EudraCT Number)
Record Dates: First submitted 2016-06-01; First posted 2016-07-07 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Relapsed/Refractory B Cell Malignancies; Mantle Cell Lymphoma and Diffuse Large B Cell Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Treatment-Naive B Cell Malignancies
Keywords: TL-895; Tyrosine Kinase Inhibitor; Lymphoma; Open; Phase I; Phase II; CLL; SLL
MeSH Terms: conditions — Recurrence; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- TL-895 80/160 mg QD in R/R Participants (Experimental): Participants received TL-895 80 mg powder in capsule (PiC) orally once daily (OD) for 3 days followed by TL-895 160 mg OD in fasted state for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 300 mg QD in R/R Participants (Experimental): Participants received TL-895 300 mg PiC orally OD in fasted state for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 600 mg QD in R/R Participants (Experimental): Participants received TL-895 600 mg PiC orally OD in fasted state for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 300 mg BID in R/R Participants (Experimental): Participants received TL-895 300 mg PiC orally twice daily (BID) in fasted state for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 900 mg QD in R/R Participants (Experimental): Participants received TL-895 900 mg PiC orally QD in fasted state for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 100 mg BID in R/R Participants (Experimental): Participants received TL-895 100 mg BID orally with food for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 150 mg BID in R/R Participants (Experimental): Participants received TL-895 150 mg BID orally with food for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 150 mg BID in Treatment Naïve Participants (Experimental): Participants received TL-895 150 mg BID orally with food for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 100 mg BID in Treatment Naïve Participants (Experimental): Participants received TL-895 100 mg BID orally with food for 28 days in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895
- TL-895 150 mg BID & navtemadlin 240mg QD in R/R Participants without 17p(del) (Experimental): Participants received navtemadlin 240 mg administered QD on Days 1-7 in combination with TL-895 150 mg BID orally with food for 28 days with in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895; Drug: Navtemadlin
- TL-895 150 mg BID & navtemadlin 240mg QD in Treatment Naïve Participants without 17p(del) (Experimental): Participants received navtemadlin 240 mg administered QD on Days 1-7 in combination with TL-895 150 mg BID orally with food for 28 days with in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895; Drug: Navtemadlin
- TL-895 150 mg BID & navtemadlin 240mg QD in R/R Participants with 17p(del) (Experimental): Participants received navtemadlin 240 mg administered QD on Days 1-7 in combination with TL-895 150 mg BID orally with food for 28 days with in each 28 day cycle until disease progression, withdrawal of consent, or discontinuation from the study.
  Interventions: Drug: TL-895; Drug: Navtemadlin

INTERVENTIONS:
Drug: TL-895 — TL-895 is an experimental tyrosine kinase inhibitor anticancer drug taken by mouth.
Drug: Navtemadlin — Navtemadlin is an experimental MDM2 anticancer drug taken by mouth.
  Arms: TL-895 150 mg BID & navtemadlin 240mg QD in R/R Participants with 17p(del); TL-895 150 mg BID & navtemadlin 240mg QD in R/R Participants without 17p(del); TL-895 150 mg BID & navtemadlin 240mg QD in Treatment Naïve Participants without 17p(del)

SUMMARY:
The purpose of this research study is to determine the safety and tolerability of TL-895. There are 2 parts of this study. Part 1 tested increasing doses of TL-895 to identify the recommended safe dose for participants with relapsed/refractory (R/R) B cell malignancies who failed at least 1 but no more than 3 prior therapies. Part 1 of this study is no longer enrolling participants.

Arms 1 & 2 of Part 2 of this study will test different doses of TL-895 in participants with R/R CLL or SLL who have failed at least 1 prior therapy. Arms 1 & 2 of Part 2 of this study is randomized (like the flip of a coin) to receive a specific treatment dose. If someone participates in arms 1 or 2 of Part 2, the dose they receive will be either 100mg twice a day or 150mg twice a day.

Arms 3 and 4 of Part 2 of this study will test the 150mg and 100mg BID dose of TL-895, respectively in treatment naïve participants with CLL/SLL.

Arms 5 and 6 of Part 2 will test 150mg TL-895 BID in combination with 240 mg navtemadlin QD in participants with relapsed/refractory and treatment naïve without 17p(del). Arm 7 will test 150mg TL-895 in combination with 240 mg navtemadlin QD in participants with relapsed/refractory CLL/SLL with 17p(del).

Every participant in this study will receive TL-895.

ELIGIBILITY:
Inclusion Criteria

* Relapsed/refractory CLL or relapsed/refractory SLL (Arms 1, 2, 5, and 7)
* Treatment naïve CLL or SLL (Arm 3, 4, and 6)
* ECOG performance status of ≤ 2
* Adequate hematologic, hepatic, and renal functions

Exclusion Criteria

* Prior treatment with any BTK or PI3K inhibitors
* History of major organ transplant
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2016-08-26 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Dose Escalation): DLTs (Dose Limiting Toxicities) during Cycle 1 | Baseline up to the end of cycle 1 (28 days)
  DLT is defined as any of the adverse event (AEs) of a certain grade or above, related to drug.
Part 2 (Dose Expansion): Overall Response Rate (ORR) | Baseline up to end of study (2 years after last patient enrolled)
  The proportion of subjects achieving CR, CRi, nodular partial response (nPR), partial response (PR), or PR with lymphocytosis (PR-L) at any time while on the study based on iwCLL response criteria (2), as assessed by investigators

SECONDARY OUTCOMES:
Part 1 (Dose Escalation): Best Overall Response (BOR)/Progression Free Survival (PFS) | Baseline up to 6 months on treatment
  Defined by the length of time during the treatment of the disease, that a participant lives with the disease but it does not get worse based on investigator assessments
Part 2 (Dose Expansion): Overall CR/CRi rate | Baseline up to end of study (2 years after last patient enrolled)
  The proportion of subjects achieving CR/CRi based on iwCLL response criteria
Part 2: Duration of Clinical Response (DOR) | Baseline up to end of study (2 years after last patient enrolled)
  Time from initial response to disease progression or death from any cause
Part 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Baseline up to end of study (2 years after last patient enrolled)
  Incidence, nature, severity of treatment-emergent adverse events (TEAEs), and deaths, including cause of death, from screening up to the end of study visit of participants with CLL/SLL who have failed at least 1 line of therapy
Part 2: Assessment of Safety and Tolerability via Clinical Measurements | Baseline up to end of study (2 years after last patient enrolled)
  Assessments including but not limited to clinical laboratory measurements, ECGs, vital signs, and ECOG performance

CONTACTS AND LOCATIONS:
Locations (17):
- United States (2):
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - The West Clinic, Germantown, Tennessee
- Hungary (2):
  - Debreceni Egyetem - Borgyógyászati Klinika, Debrecen
  - Eger Markhot Ferenc Kórház, Eger
- Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi - Istituto di Ematologia e Oncologia Medica, Bologna, Italy
- Poland (5):
  - Examen sp. z o. o., Skorzewo, Poznań
  - Pratia MCM Krakow, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im sw Jana z Dukli Oddzial Hematologiczny, Lublin
  - Szpital Wojewódzki, Opole
  - Nasz Lekarz Przychodnie Medyczne, Torun
- Russia (2):
  - Saint Petersburg State Medical University, Saint Petersburg
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
- Ukraine (3):
  - Communal Non-profit Enterprise Regional Center of Oncology, Kharkiv
  - Kyiv City Clinical Hospital #4, Kyiv
  - Mykolaiv Regional Clinical Hospital, Mykolaiv
- United Kingdom (2):
  - University College London Hospitals - NIHR/Wellcome Trust, London
  - Derriford Hospital - Dept of Haematology, Plymouth

REFERENCES:
- [Background] Eugenio Gaudio, Chiara Tarantelli, Emanuele Zucca, Davide Rossi, Anastasios Stathis, Francesco Bertoni. The two novel BTK-inhibitors M2951 and M7583 show in vivo anti-tumor activity in pre-clinical models of B cell lymphoma [abstract]. In: Proceedings of the American Association for Cancer Research Annual Meeting 2017; 2017 Apr 1-5; Washington, DC. Philadelphia (PA): AACR; Cancer Res 2017;77(13 Suppl):Abstract nr 4182. doi:10.1158/1538-7445.AM2017-4182
- [Background] Goodstal SM, Lin J, Crandall T, Crowley L, Bender AT, Pereira A, Soloviev M, Wesolowski JS, Iadevaia R, Schelhorn SE, Ross E, Morandi F, Ma J, Clark A. Preclinical evidence for the effective use of TL-895, a highly selective and potent second-generation BTK inhibitor, for the treatment of B-cell malignancies. Sci Rep. 2023 Nov 21;13(1):20412. doi: 10.1038/s41598-023-47735-z. PMID 37989777
- [Background] Wojciech Jurczak, Simon Rule, William Townsend, David Tucker, Martin Dyroff, Barbara Sarholz, Jürgen Scheele, John G. Gribben and Pier Luigi Zinzani. First in Human, Phase I/II Trial of the Bruton's Tyrosine Kinase Inhibitor (BTKi) M7583 in Patients with B Cell Malignancies: Study Design and Initial Outcomes. Blood 2017 130:2778.
- [Background] Jurczak W, Rule S, Townsend W, Tucker D, Sarholz B, Scheele J, Dyroff M, Gribben JG, Dlugosz-Danecka M, Zinzani PL. Phase I, first-in-human trial of Bruton's tyrosine kinase inhibitor M7583 in patients with B-cell malignancies. Leuk Lymphoma. 2021 Oct;62(10):2392-2399. doi: 10.1080/10428194.2021.1913139. Epub 2021 Apr 24. PMID 33896333